CLINICAL TRIAL: NCT07396285
Title: UCSF Center for Genome Surgery Biobank and Registry
Status: Not yet recruiting | Type: Observational
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Other Study IDs: UCSF_CGS_Biobank_Registry
Record Dates: First submitted 2025-10-07; First posted 2026-02-09 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Any Conditions That Are Genetic or Suspected to be Genetic in Origin
Keywords: Genetic; gene therapy

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Center for Genome Surgery Case Series Discussion
- Enrollment in Registry and Biobank

SUMMARY:
Gene editing approaches (including but not limited to: CRISPR, LNP, AAV, RNAi etc.) for the medical specialty of interventional genomics require (1) determination of the clinical relevance of genomic variants and (2) systematic evaluation of the 'editability' of those variants. Here, we seek to use in silico and in vitro analyses of genomic, cellular, and clinical data/specimens to (1) identify novel pathogenic variants underlying diseases and (2) examine the specificity and efficacy of various gene editing components across the entire human genomic landscape.

ELIGIBILITY:
Inclusion Criteria:

For initial screening and discussion at huddle call:

* Male and female individuals of any age, including pregnant women and their fetuses at any gestational age.
* Self-referred or referred through their provider to the UCSF Center for Genome surgery/Interventional Genomics Board for a condition that is genetic or suspected to be genetic in origin.
* UCSF patient OR consents to allow for their case to be presented at the IGB huddle.

For enrollment into registry or biobanking:

* Any above participant that the IGB agrees would be appropriate for enrollment in the registry and biobanking portion of this protocol OR Any male or female family member of any age of someone enrolled in the registry and biobanking portion of this protocol.
* Provides informed consent for participation in the registry and biobanking portion of the protocol.

Exclusion Criteria:

For initial screening and discussion at huddle call:

* Individuals who have previously been discussed by the IGB and determined to not be appropriate to move forward into the registry and biobanking portion of the protocol, unless new information related to their case may change the initial assessment.
* Individuals who are not impacted by a genetic or suspected genetic condition.

For enrollment into registry or biobanking:

-Any participant that the IGB agrees is inappropriate for enrollment in the registry and biobanking portion of this protocol.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Any individual diagnosed with a genetic disorder that may be amenable to gene therapy.
Sampling Method: Non-Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2026-05-01 (Estimated); Primary Completion 2050-12 (Estimated); Study Completion 2050-12 (Estimated)

PRIMARY OUTCOMES:
Improve our understanding of how specific mutations lead to dysfunction and cause disease | Up to 25 years
Empirically assess the edibility of individual participant genomic variants in silico and in patient-derived cells for the purpose of bespoke genomic therapies. | Up to 25 years

OTHER OUTCOMES:
Support preclinical investigations of gene therapies specific to participants | Up to 25 years

CONTACTS AND LOCATIONS:
Overall Officials: Tippi Mackenzie, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified specimens and data may be shared with other researchers

REFERENCES:
- [Background] Tsai, S., Zheng, Z., Nguyen, N. et al. GUIDE-seq enables genome-wide profiling of off-target cleavage by CRISPR-Cas nucleases. Nat Biotechnol 33, 187-197 (2015). https://doi.org/10.1038/nbt.3117
- [Background] Lazzarotto, C.R., Malinin, N.L., Li, Y. et al. CHANGE-seq reveals genetic and epigenetic effects on CRISPR-Cas9 genome-wide activity. Nat Biotechnol 38, 1317-1327 (2020). https://doi.org/10.1038/s41587-020-0555-7
- [Background] Ioannidis, N. M., Rothstein, J. H., Pejaver, V., Middha, S., McDonnell, S. K., Baheti, S., Musolf, A., Li, Q., Holzinger, E., Karyadi, D., Cannon-Albright, L. A., Teerlink, C. C., Stanford, J. L., Isaacs, W. B., Xu, J., Cooney, K. A., Lange, E. M., Schleutker, J., Carpten, J. D., Powell, I. J., … Sieh, W. (2016). REVEL: An Ensemble Method for Predicting the Pathogenicity of Rare Missense Variants. American journal of human genetics, 99(4), 877-885. https://doi.org/10.1016/j.ajhg.2016.08.016